CLINICAL TRIAL: NCT06013488
Title: A Character-Strengths Based Coaching Program for Rural Community Health Workers to Address Their Work Stress in India: Protocol for a Two-arm Randomized Controlled Trial
Brief Title: Character-Strengths Based Coaching For Work-Stress Reduction For Health Workers
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Templeton World Charity Foundation (Other)
Responsible Party: Principal Investigator, Anant Bhan, Principal Investigator, Sangath
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: TWCF0635
Record Dates: First submitted 2023-08-22; First posted 2023-08-28 (Actual); Last update posted 2024-11-20 (Actual); Status verified 2024-11

CONDITIONS: Work Related Stress; Burnout, Psychological; Mental Health Issue
Keywords: character strengths; community health workers; work stress; India; randomized controlled trial; positive psychology
MeSH Terms: conditions — Occupational Stress; Burnout, Psychological

STUDY DESIGN:
Intervention Model Description: This study employs a 2-arm parallel randomized controlled trial design. Participants will be randomly allocated to 1) a character-strengths based coaching intervention consisting of a five-day residential workshop and supplemental 8- to 10-week remote telephonic coaching support in addition to 'routine (health system) supervision' (face-to-face by a supervisor in groups of 1 supervisor for ~20 health workers), or 2) 'routine supervision' alone.
Who Masked: Outcomes Assessor
Masking Description: In this trial, the Outcome Assessors administering study assessments at baseline and at 1-, 3- and 6-month follow-up will be masked to the intervention arm that participants are allocated to receive. Masking outcome assessors will minimize potential bias due to knowledge of which arm the participant is allocated to, and can ensure unbiased ascertainment of study outcomes. For allocation concealment, the intervention allocation for each participant will not be revealed to the participant until they have been enrolled into the trial, to avoid selection bias.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Arm (Experimental): Participants (health workers) allocated to this arm continue to receive the traditional weekly supervision delivered by their supervisor, assigned by the health system, in a face-to-face mode in groups of 1:20 (1 supervisor for a group of ~20 health workers). In addition, participants receive a 5-day residential coaching workshop involving character-strengths based strategies to reduce work-stress, followed by supplemental 8- to 10-week remote telephonic coaching support, after the workshop when they resume work (and experience stressors). The weekly coaching support calls typically last for 30-45 minutes and are delivered by an assigned intervention coach (by the study team) to the health worker (1:1).
  Interventions: Behavioral: Character Strengths Based Coaching Support; Behavioral: Routine Supervision
- Control Arm (Active Comparator): Participants (health workers) allocated to this arm receive the traditional weekly supervision delivered by their supervisor, assigned by the health system, in a face-to-face mode in groups of 1:20 (1 supervisor for a group of ~20 health workers).
  Interventions: Behavioral: Routine Supervision

INTERVENTIONS:
Behavioral: Character Strengths Based Coaching Support — Residential (five day) workshop and remote (weekly) telephonic support for 8 to 10 weeks
  Arms: Intervention Arm
Behavioral: Routine Supervision — Weekly face-to-face supervision by supervisor in groups of ~20 (1 supervisor for ~20 health workers)

SUMMARY:
The purpose of this two-arm, parallel group individual randomized controlled trial is to evaluate the effectiveness of a character-strengths based coaching intervention consisting of a five-day residential workshop focusing on the use of character-strengths to address work-stress in routine situations supplemented by 8- to 10-week remote telephonic weekly coaching sessions to support rural health workers, as they face stressful situations and apply the strategies learnt in the workshop. The arms are: the character-strengths based intervention added to routine health worker supervision (weekly, by the supervisor) and routine supervision alone (control arm). The target sample comprises 330 government contracted 'ASHAs' (rural resident women, lay health workers) in the Sehore district of Madhya Pradesh, one of the most populous and poorest of the states in India. Scores on the 'Authentic Happiness Inventory (AHI)' will serve as the primary outcome for self-reported wellbeing and will be compared between arms at 3-month follow-up. Secondary ASHA-level outcomes will include assessment of self-reported affect, self-efficacy, flourishing, burnout, and motivation. We will also collect exploratory outcomes, including routine service delivery indicators to assess any effect of changes in well-being on ASHA's regular work performance, and resulting patient-level outcomes like satisfaction with services, and depression severity levels after receiving community-based depression care delivered by the ASHAs. We will also evaluate the costs of delivering the intervention and those incurred by ASHAs due to their participation in the intervention. Assessors blind to participant allocation will collect outcomes at baseline, 1-month and 3-month follow-up, as well as at 6-month follow-up, to ascertain differences in outcomes between arms. In addition, scores of ASHAs' self-perceived character strengths will be collected at baseline and 3-month follow-up as exploratory variables.

DETAILED DESCRIPTION:
Character strengths-based interventions are found to be effective in improving well-being and reducing burnout amongst healthcare workers. But there is scarce knowledge on the use of structured positive psychology interventions for reduced work-stress and improving mental wellbeing of Accredited Social Health Activists (ASHAs). ASHAs are village level community lay health care workers who provide the bulk of the health care services in rural India. ASHAs are overworked and underpaid and subjected to considerable stress for both professional and domestic reasons (being married, rural, traditional women). This study will test the effectiveness of a 'character-strengths' based coaching intervention on ASHAs' self-reported wellbeing.

This study will evaluate the effectiveness of the aforementioned coaching intervention compared with routine supervision (delivered by one ASHA supervisor, weekly, face-to-face, typically in groups of ~20 ASHAs) on self-reported wellbeing score at 3-month follow-up. In this trial, a total of 330 ASHAs will be recruited in Sehore District of Madhya Pradesh, a large and predominantly rural state situated in central India.

The development of the coaching intervention (published elsewhere, Khan A et al., 2023) involved: (1) formative work, (2) blueprint development, (3) content development, (4) content-testing, and focus groups discussions to evaluate the feasibility and acceptability of the intervention, specifically the coaching workshop. This was followed by thematic qualitative analysis of ASHA perspectives/feedback to inform further modifications to the workshop. Intervention development occurred over 11 months, and the final coaching material consisted of a 'content manual' (for ASHAs) with four modules including character-strengths based 'strategies' to address challenges/stressors arising at health facilities, village communities and homes. Coaching material also included a workshop 'facilitator's manual' having session-wise detailed instructions, a list of 'energizers' and plans for the coaching workshop; and a protocol for remote telephonic coaching support to provide follow-on weekly support to ASHAs (typically 30-45 minute phone-calls) as they resume work (and experience stressors) and reinforce the learnings of the workshop.

This trial will determine whether character-strengths based coaching is an effective and scalable approach for reducing work-stress and improving mental wellbeing of rural ASHAs in low-resource settings. The findings from this trial will inform broader efforts to develop similar stress-reduction interventions, which are necessary for related cadres (e.g., nurse midwives, rural doctors) in low-resource settings in India and other low- and middle-income countries.

ELIGIBILITY:
Inclusion Criteria:

* All rural ASHAs residing and working in Sehore district, Madhya Pradesh (verified in the health system records) and who have been trained by the study team on delivering community-based depression care

Exclusion Criteria:

* ASHAs who plan to migrate within six months of recruitment
* ASHAs who do not plan to continue working, or those who have resigned or planning to change jobs within six months of recruitment
* ASHAs with urban catchment areas
* ASHA supervisors will not be included owing to hierarchical differences in these two cadres and their potential effects on absorption of intervention content, and thereby on their wellbeing (primary outcome of interest)
* ASHAs who have difficulties in using a smartphone

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 330 (Estimated)
Dates: Start 2023-08-21 (Actual); Primary Completion 2025-07-30 (Estimated); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
Mean score on the Authentic Happiness Inventory (AHI) | Baseline, 3-month and 6-month follow-up
  Authentic Happiness Inventory (AHI) is a subjective measure for the assessment of happiness. We have used the term 'wellbeing' in the protocol to represent this specific measure of happiness. AHI includes 24 sets of five statements [e.g., ranging from 1 ("I feel like a failure") to 5 ("I feel I am extraordinarily successful")] from which, the respondent chooses the statement that best describes her feelings in the past one week. AHI has been designed for monitoring upward changes in happiness and has often been used in positive psychology intervention studies. Internal consistency at pre-test has been reported to be high (Cronbach's α = 0.94). AHI will be administered at baseline, and at 3 and 6 months thereafter. The primary outcome analysis will involve a comparison of mean AHI scores between arms at 3-month follow-up.

SECONDARY OUTCOMES:
Mean score on the Positive and Negative Affect Schedule (PANAS) | Baseline, 1-month and 3-month follow-up
  The 10-item international Positive and Negative Affect Schedule (PANAS) Short Form (I-PANAS-SF) will be used to assess ASHA affect due to its acceptable psychometric properties such as cross-cultural stability and factorial invariance. ASHA's affect will be assessed as a mediating variable to examine its potential role in affecting wellbeing (AHI score).
Mean score on Flourish Index (FI) and Secure Flourish Index (SFI) | Baseline, 1-month and 3-month follow-up
  The "Flourish" index (FI) consists of two questions from each of the following domains: happiness and life satisfaction, mental and physical health, meaning and purpose, character and virtue, and close social relationships. Each question is assessed on a scale of 0 - 10. FI score is obtained by adding the scores from each of these ten questions (total: 0-100). The "Secure Flourish" index (SFI) is similar to the FI, except for two additional questions on financial and material stability, which may indicate the capacity to sustain flourishing across the aforesaid domains. The FI and SFI scores are reported as averages of the questions (rather than sums), therefore all scores are scaled from 0-10. Studies have put forth Cronbach's α = 0.89 for FI and Cronbach's α = 0.86 for SFI. FI and SFI will be assessed as mediating variables for their potential effects on wellbeing.
Mean score on Occupational Self-Efficacy Scale (OSES) | Baseline, 1-month and 3-month follow-up
  We are using the Occupational Self Efficacy Scale (OSES) given that its psychometric properties have been analyzed in the Indian context, and to that extent, we will adapt the scale among ASHAs for making any linguistic modifications. Self-efficacy will also be assessed as a mediating variable for its potential effect on wellbeing.
Mean score on the Emotional exhaustion sub-scale of the Maslach Burnout Inventory-Human Service Survey (MBI-HSS) | Baseline, 3-month and 6-month follow-up
  This tool is designed to measure burnout in professionals working in the human services. The overall questionnaire measures three burnout components: emotional exhaustion (8 items, Cronbach's α = 0.89), depersonalization (5 items, Cronbach's α = 0.69) and reduced personal accomplishment (7 items, Cronbach's α = 0.79). Emotional exhaustion is seen as the core component of this tool. Items are scored on a seven-point Likert's style scale. We will assess burnout as an extrinsic outcome variable i.e., potentially affected by the aforementioned mediator variables.
Mean score on the motivation scale for Indian frontline workers | Baseline, 3-month and 6-month follow-up
  We are using the tool pretested by Tripathy et al for Indian frontline health workers (including ASHAs, Auxiliary Nurse Midwives and Aanganwadi Workers) adapted from a motivation construct developed by Mbindyo et al, which was adapted from Bennet et al. Like burnout, we will assess motivation as an extrinsic outcome variable.

OTHER OUTCOMES:
Service delivery indicators | Baseline, 1-month, 3-month and 6-month follow-up
  ASHAs' routine service delivery indicators will be gathered from the block (sub-district unit) administration office. Examples of these indicators include proportion of antenatal and postnatal home visits completed (out of those expected) and proportion of eligible infants and children who were immunized. The study hypothesizes a secondary effect of improvement in ASHA's mental wellbeing on the delivery of her services. Indicators will be descriptively compared between arms. Indicators related to delivery of community-based mental health care such as number of sessions delivered for brief psychological treatment of people identified with depression, will also be compared between arms.
Healthy Activity Program (HAP) session quality | 3-month and 6-month follow-up
  As part of this trial, all enrolled ASHAs (both arms) are required to undergo training in the delivery of community based brief psychological treatment for depression (HAP). The digital HAP training model has been published previously (Naslund et al., 2021; NCT04157816). HAP typically includes weekly sessions for 6-8 weeks at the patient's home/mutually agreed location between the patient and the ASHA (village-level). HAP sessions will be rated using the 20-item Quality of Healthy Activity Program rating scale (Q-HAP) assessing treatment-specific and general therapy skills. ASHAs will record their sessions using their smartphones and the audio files will be sent to the HAP supervisors following all ethical procedures. Scores of the available rated sessions will be compared between arms at predetermined time-points.
Patient satisfaction with HAP | 3-month follow-up of the patient receiving HAP by ASHA
  All HAP-trained ASHAs will start screening adult individuals in their respective villages for depression using the nine-item Patient Health Questionnaire (PHQ-9). Individuals screened positive (PHQ-9 score >=10) will be approached by the study team for consent to participate in the study. After consent, the research team member will administer a baseline social and demographic assessment and retrieve the PHQ-9 score as the 'baseline' for record purposes, and the ASHA will start delivering the HAP sessions. After 3 months (from baseline), the research team will visit the patient to assess their satisfaction with HAP using the eighteen item Patient Satisfaction Questionnaire (PSQ-18) to measure the general satisfaction, technical quality, interpersonal aspects, communication, accessibility and convenience. Higher value of the composite score indicates more satisfaction.
Remission on nine-item Patient Health Questionnaire (PHQ-9) | 3-month follow-up of the patient receiving HAP by ASHA
  All patients receiving HAP by respective ASHAs will be approached for endpoint assessment of PHQ-9 score (by research team member), 3 months after assessment of their baseline score (as screened by the ASHA). The study hypothesizes a linkage between improved mental wellbeing of ASHAs and resulting improvements in service delivery, and patient satisfaction and patient clinical outcomes. Remission at endpoint is defined by a follow-up PHQ-9 score of <5.
Cost assessment of the character-strengths based coaching intervention | Day-5 of residential workshop and 2nd, 4th, 6th and 8th coaching support call (only for intervention arm ASHAs)
  ASHAs allocated to the intervention arm will receive a cost survey to estimate their expenses during the 5-day residential coaching workshop and their time/effort put on the workshop and 8- to 10-week (weekly) remote telephonic coaching support. The cost survey for the workshop will be delivered on day-5 of the workshop by the intervention team and the cost survey for remote coaching will be delivered at the end of 2nd, 4th, 6th and 8th coaching call.
Self-perceived strengths assessment | Baseline and 3-month follow-up
  The Self-Perceived Strengths (SPS) scale, is a brief 24-item self-administered vignette-based measure of character strengths developed and validated for the Indian population (Tripathi et al., 2015). The 24 items have the six-point Likert-type rating (responses ranging from "very different from me" (1) to "very much like me" (6)). Each vignette describes a hypothetical individual having the cognitive and behavioral characteristics of a particular character strength, without specifying the name of the strength. Participants are required to specify the degree of similarity-dissimilarity ("very different from me"-> "very much like me") with the hypothetical person. Test-retest reliability ranges between 0.43-0.8 and strength coefficients are reported to be significant at 0.01 level. We will assess the change in the self-reported strengths expression from baseline to follow-up, compared between arms.

CONTACTS AND LOCATIONS:
Overall Officials: Anant Bhan, Principal Investigator — Site Head, Sangath Bhopal Hub
Locations (1):
- Sangath Bhopal Hub, Bhopal, Madhya Pradesh, India

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Khan, A., Sharma, L., Agrawal, S. et al. Development of a character-strengths based coaching program for rural community health workers to address their work stress in Madhya Pradesh, India. Curr Psychol (2023). https://doi.org/10.1007/s12144-023-04673-3